CLINICAL TRIAL: NCT00470093
Title: A Pilot Study of Differentiation Therapy in Multiple Myeloma Using Interleukin-6 and Interferon-a
Brief Title: Interferon Alfa and Interleukin-6 in Treating Patients With Recurrent Multiple Myeloma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0620; P30CA006973 (NIH); P01CA015396 (NIH); NA_00002178 (Other: JHMIRB)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Interleukin-6

ARMS (1):
- Interleukin-6 and Interferon-α (Experimental): Subjects will be started on recombinant interferon-α at a dose of 3 million units SQ daily, escalating the dose by 1 million units every week as tolerated to a maximum dose of 3 million units/m2/day. Following a minimum of one month of interferon therapy with two weeks on a stable dose, subjects will begin recombinant interleukin-6 therapy at a dose of 2.5 ug/kg/day.
  Interventions: Biological: recombinant interferon-α; Biological: recombinant interleukin-6

INTERVENTIONS:
Biological: recombinant interferon-α
Biological: recombinant interleukin-6

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells. Interleukin-6 may stimulate the white blood cells to kill cancer cells. Giving interferon alfa together with interleukin-6 may kill more cancer cells.

PURPOSE: This clinical trial is studying the side effects and how well giving interferon alfa together with interleukin-6 works in treating patients with recurrent multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with recurrent multiple myeloma treated with recombinant interferon alfa and recombinant interleukin-6.
* Determine the safety and optimal dose of this regimen in these patients.
* Determine the toxicity of this regimen in these patients.
* Determine the impact of this regimen on clonogenic growth of myeloma cells in serial in vitro assays.

OUTLINE: This is a pilot study.

Patients receive recombinant interferon alfa subcutaneously (SC) once daily. Beginning 1 month later, patients also receive recombinant interleukin-6 SC once daily. Treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of recurrent multiple myeloma
* Must have received ≥ 2 prior therapies

PATIENT CHARACTERISTICS:

* Performance status 0-3

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Huff, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was a screen failure.
Groups:
- Interleukin-6 and Interferon-α: Subjects will be started on recombinant interferon-α at a dose of 3 million units SQ daily, escalating the dose by 1 million units every week as tolerated to a maximum dose of 3 million units/m2/day. Following a minimum of one month of interferon therapy with two weeks on a stable dose, subjects will begin recombinant interleukin-6 therapy at a dose of 2.5 ug/kg/day.
  recombinant interferon-α
  recombinant interleukin-6
Period: Overall Study
Arm/Group | Interleukin-6 and Interferon-α
Started | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Interleukin-6 and Interferon-α
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 54.5 [50 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate as Assessed by Number of Participants With Partial or Complete Response by Bladé Criteria.
Description: Number of participants with partial or complete response by Bladé criteria where partial response is defined as a >= 50% decrease in serum paraprotein or 90% decrease in urinary light chains (for participants without measurable serum paraprotein). Complete response is defined as negative serum and urine immunofixation and a bone marrow aspirate with < 5% plasma cells.
Time Frame: Up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Interleukin-6 and Interferon-α
Number analyzed (Participants) | 2
Participants | 0

2. Primary Outcome: Toxicity as Measured by Number of Participants Who Discontinued Treatment Due to Adverse Events
Description: Number of participants who discontinued the protocol due to adverse events.
Time Frame: Up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Interleukin-6 and Interferon-α
Number analyzed (Participants) | 2
Participants | 2

3. Primary Outcome: Optimal Dose of Interleukin-6
Description: Maximum tolerated dose found using a standard 3+3 dose escalation model.
Time Frame: Up to 5 months
Population: This outcome cannot be evaluated as zero participants tolerated the study regimen. All participants were enrolled on the 2.5 mg arm and a maximum tolerated dose was not found.
Arm/Group | Interleukin-6 and Interferon-α
Number analyzed (Participants) | 0

4. Primary Outcome: Impact of Treatment on Growth of Myeloma Cells
Description: Percentage change in growth of in vitro myeloma cells from baseline to end of study.
Time Frame: Day 0, Day 14, Months 1, 2, 4, and 6 of combined therapy, and end of study
Population: Zero participants tolerated protocol therapy and the research sample blood draws were therefore not completed as planned. Because of this, the data from this outcome could not be collected.
Arm/Group | Interleukin-6 and Interferon-α
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 5 months
Description: Adverse events were assessed every two weeks through the first two months of combination therapy, then monthly through the end of the study.
Arm/Group | Interleukin-6 and Interferon-α
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interleukin-6 and Interferon-α (N=2)
Cold-like symptoms (General disorders) | 2 (2)
Anorexia (General disorders) | 2 (4)
Fever (General disorders) | 2 (3)
Chills (General disorders) | 2 (4)
Diaphoresis (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Excessive sleepiness (General disorders) | 1 (1)
Flu-like symptoms (General disorders) | 2 (2)
Weight loss (General disorders) | 1 (1)
Xerostomia (Skin and subcutaneous tissue disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Anemia (Investigations) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 2 (4)
Confusion (Nervous system disorders) | 2 (3)
Dizziness (Nervous system disorders) | 2 (4)
Memory loss (Nervous system disorders) | 2 (3)
Headache (General disorders) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain - neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Voice changes (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Salt sensitivity (Immune system disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Constipation (General disorders) | 1 (1)
Depression (Nervous system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No